CLINICAL TRIAL: NCT02423473
Title: Composite Resin Plus Connective Tissue Graft to Treat Gingival Recession Associated With Non-carious Cervical Lesion. Randomized Clinical Trial
Brief Title: Composite Resin Plus Connective Tissue Graft.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 071/2010
Record Dates: First submitted 2015-04-03; First posted 2015-04-22 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Filtek Supreme

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Connective tissue graft (CTG) (Active Comparator): After local anesthesia, the surgical procedure performed was the trapezoidal-type of CAF (de Sanctis & Zucchelli, 2007). After the flap was raised, the exposed root surface was gently scaled and planed until it became smooth. Afterward, a thin and small connective tissue graft that was sutured over the root surface. Then, the flap was coronally positioned and sutured to completely cover the graft.
  Interventions: Procedure: Connective tissue graft
- Connective tissue graft plus composite resin restoration. (Experimental): After local anesthesia, the surgical procedure performed was the trapezoidal-type of CAF (de Sanctis & Zucchelli, 2007). After the flap was raised, a sterile rubber dam was placed to isolate the operative field and the non-carious cervical lesion restoration was performed with a nanocomposite resin (Filtek Supreme - 3M ESPE - St. Paul, MN, USA), following the manufacturer's instructions. Afterward, a thin and small connective tissue graft that was sutured over the restoration surface. Then, the flap was coronally positioned and sutured to completely cover the graft.
  Interventions: Procedure: Connective tissue graft; Procedure: Composite resin restoration (Filtek Supreme - 3M)

INTERVENTIONS:
Procedure: Connective tissue graft — Periodontal surgical technique to treat gingival recessions
  Other Names: Periodontal plastic surgery
Procedure: Composite resin restoration (Filtek Supreme - 3M) — Restorative procedure do treat tooth structure loss
  Other Names: Non-carious cervical lesion restoration
  Arms: Connective tissue graft plus composite resin restoration.

SUMMARY:
The aim of the present study is to evaluate the clinical, aesthetic and patient-centered parameters of connective tissue graft associated or not with composite resin for the treatment of gingival recession.

DETAILED DESCRIPTION:
This was a prospective, parallel and controlled clinical trial.

Group CTG (n = 18) - patients who received connective tissue graft to treat gingival recession associated with non-carious cervical lesion. Group CTG+RC (n = 18) - patients who received connective tissue graft plus resin composite restoration to treat gingival recession associated with non-carious cervical lesion.

The surgeries, as well as all postoperative follow-up, were performed at the dental clinic of ICT- UNESP. Two horizontal incisions were made at right angles to the adjacent interdental papillae, without interfering with the gingival margins of neighboring teeth. Two oblique vertical incisions were extended beyond the mucogingival junction, and a trapezoidal mucoperiosteal flap was raised up to the mucogingival junction. After this point, a split-thickness flap was extended apically, releasing the tension and favoring coronal positioning of the flap.The exposed root surface was gently scaled and planed until it became smooth in the CTG group. For those allocated to CTG+RC group, a sterile rubber dam was placed to isolate the operative field and the non-carious cervical lesion restoration was performed with a nanocomposite resin (Filtek Supreme - 3M ESPE - St. Paul, MN, USA), following the manufacturer's instructions. Afterward, the both groups received a thin and small connective tissue graft that was sutured over the root/restoration surface. Then, the flap was coronally positioned and sutured to completely cover the graft.

Clinical parameters were assessed at baseline and 3 and 6 months post-operatively.

Statistical Analysis The null hypothesis considered in the study was the absence of difference in the clinical parameters between the different groups. For data analysis, the statistical program was used (Sigmaplot). The demographic and clinical data were compared between the groups using Student's t-test. The data were first analyzed for homogeneity using the Shapiro-Wilk test, which indicated non-normal distribution. . Those presenting Shapiro-Wilk p values < 0.05 were analyzed using a Friedman test (for intragroup comparisons) and Mann-Whitney tests (for intergroup comparisons). Patients' esthetics and discomfort measures using VAS were analyzed by T-tests. The frequency of sites that were scored as very good or excellent in each group by QCE analysis, the frequency of complete root coverage, BOP, and the presence or absence of plaque at the site were compared using χ2 tests. Intergroup RES comparisons were performed with a T-test. A significance level of 0.05 was adopted.

ELIGIBILITY:
Inclusion Criteria:

* presenting Miller class I or II gingival recession in the maxillary canines or premolars associated with non-carious cervical lesion;
* teeth included in the study should present pulp vitality;
* patients presenting no signs of active periodontal disease and full-mouth plaque and bleeding score ≤ 20%;
* patients older than 18 years old;
* probing depth ˂ 3 mm in the included teeth;
* patients who agreed to participate and signed an informed consent form

Exclusion Criteria:

* patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, and diabetes, among others) that will contraindicate the surgical procedure
* patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure
* smokers or pregnant women
* patients who underwent periodontal surgery in the area of interest; and

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Percentage of defect coverage | 1 year

SECONDARY OUTCOMES:
Root coverage esthetic score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT-UNESP

REFERENCES:
- [Background] Santamaria MP, da Silva Feitosa D, Casati MZ, Nociti FH Jr, Sallum AW, Sallum EA. Randomized controlled clinical trial evaluating connective tissue graft plus resin-modified glass ionomer restoration for the treatment of gingival recession associated with non-carious cervical lesion: 2-year follow-up. J Periodontol. 2013 Sep;84(9):e1-8. doi: 10.1902/jop.2013.120447. Epub 2013 Jan 31. PMID 23368948